CLINICAL TRIAL: NCT06985745
Title: An Emulsion 2-Week Wash-out, 4-Week Application and Relapse for 2-Week Anti-acne Efficacy Clinical Study
Brief Title: Emulsion 8-Week Anti-acne Efficacy Clinical Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ChinaNorm (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C25005028
Record Dates: First submitted 2025-05-15; First posted 2025-05-22 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Female; Male; Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Group Emulsion (Other)
  Interventions: Other: Standard Cleanser, Investigational emulsion, Standard moisturizer, Standard Sunscreen

INTERVENTIONS:
Other: Standard Cleanser, Investigational emulsion, Standard moisturizer, Standard Sunscreen — Products Application and Usage Instruction:
  Wash out: T-2W ~ T0
  Frequency:
  AM: Standard cleanser + standard moisturizer + standard sunscreen PM: Standard cleanser + standard moisturizer Caution: All the products should be applied to full face. No any other skincare or facial make up products are used except provide products.
  b. Mode of application : 4-week Treatment T0 ~ T4W
  Frequency:
  AM: Standard cleanser + test emulsion (FLA#2039180 68) + standard sunscreen PM: Standard cleanser + test emulsion (FLA#2039180 68) Caution: All the products should be applied to full face. No other skincare or facial make up products are used except provide products.
  c. Mode of application : 2-week relapse T4W ~ T6W AM: Standard cleanser + standard moisturizer + standard sunscreen PM: Standard cleanser + standard moisturizer
  Usage Instruction： Test emulsion (FLA#2039180 68): Self-application 0.6 ml for full face by hand every day (2x/day).

SUMMARY:
65 male and female adult subjects will be enrolled in the study, recruited according to inclusion and non-inclusion criteria listed below, at least 60 subjects should complete questionnaire, at least 40 of them should complete clinical assessment, instrumental measurement and image capture. 20 of them should complete lipid sample collection, and at least 30 of them should complete the RCM captured.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese man and women aged from 20-40 years old.
2. Acne prone skin with combination to oil and oil skin type.
3. At least 50% self-declared sensitive skin.
4. Presenting with mild to moderate IGA (Acne Severity 0-4 scale, 2-3 score). 1) At least 5 inflammatory acne lesions (papules, pustules) on the global face. 2) At least 10 non-inflammatory acne lesions (blackhead, whitehead) on the global face.
5. Presenting with Cheek Sebaceous Pores (Skin aging ATLAS Vol.2 Asian Type) ≥ 3 score (0-5 scale)
6. At least 1 active inflammatory lesion can be tracked.
7. Subjects with acne red mark (PIE)
8. Presenting with skin lack of smoothness, radiance, brightness, softness evaluated by dermatologist and have skin redness concerns.

1) Skin smoothness (0-9 scale, 3≤ grade≤ 6) 2) Skin radiance (0-9 scale, 3≤ grade≤ 6) 3) Skin brightness (0-9 scale, 3≤ grade≤ 6) 4) Skin softness (0-9 scale, 3≤ grade≤ 6) 5) Skin redness (0-9 scale, 3≤ grade≤ 6) 9.No disagreement of dermatologist because of other reasons that exclude the participation of the subject.

10.In general good health at the time of the study. 11.Willing and able to participate as evidenced by signing of informed consent and photo release form.

12.Must be willing to comply with all study protocol requirements

Exclusion Criteria:

1. Pregnant or breast-feeding woman or woman planning pregnancy during the study. (applicable only to female)
2. With facial hair that may interfere with the assessment or image captured of the test area (applicable only to males);
3. Unable to participate in the trial according to the study schedule or other situations that are unsuitable for participation (e.g. Subject deprived of rights by a court or administrative order. Major subject to a guardianship order. Subject residing in a health or social care establishment. Patient in an emergency setting.)
4. Subject with a skin disease in the test areas (particularly e.g, acne, rosacea, eczema).
5. Subjects with history of atopy, allergic reactions, irritation or intense discomfort feelings to topical-use products, medication, cosmetic or personal care products or ingredients.
6. Subject presenting a stable or progressive serious disease (per investigator's assessment).
7. Immuno-compromised subject.
8. Subject presenting excessive exposure to sunlight or UV radiation (investigator's assessment).
9. Subjects regularly practicing aquatic or nautical sports.
10. Subjects regularly attending a sauna.
11. Subject with cardiovascular or circulatory history.
12. Subject with a history of skin cancer or malignant melanoma.
13. Anti-aging medical beauty project or anti-aging cosmetics clinical research in the last 6 months before study.
14. Participants who took oral isotretinoin capsules within the 6 months prior to the testing period.
15. Intake of antihistamines, antibiotics, corticosteroids, non-steroidal anti-inflammatories or immune-suppressants in the last 6 months before study.
16. Participants who are currently or have participated in other clinical trials within the past month.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2025-03-08 (Actual); Primary Completion 2025-05-27 (Estimated); Study Completion 2025-05-27 (Estimated)

PRIMARY OUTCOMES:
Clinical scoring for Counting of Acne | Timepoint 2Week before baseline，Baseline, Time point at 1Week , Time point at 4Week, Time point at 5Week, Time point at 6Week.
  Clinical scoring for counting of acne lesions (inflammatory, non-inflammatory, and total), acne severity IGA, and post-inflammatory erythema (PIE) count will be performed by a dermatologist on the global face area. The IGA (Investigator's Global Assessment for acne severity) is rated on a 5-point scale (0 = clear, 4 = severe), as defined in the protocol. PIE is recorded as a numeric count of red marks. Acne lesions (papules, pustules, blackheads, whiteheads) are counted individually.
Clinical scoring for Redness around acne | Baseline，Time point immediate, Time point at 1Day, Time point at 3Day, Time point at 1Week , Time point at 4Week, Time point at 5Week, Time point at 6Week.
  Clinical scoring for redness around acne will be performed by a dermatologist using a visual scale from 0 to 9, where 0 = no redness and 9 = intense redness, as defined in the protocol. Half-point scores (e.g., 0.5) may be used.
Clinical scoring for Diameter of tracking one Acne | Baseline，Time point immediate, Time point at 1Day, Time point at 3Day, Time point at 1Week.
  The measurement of the diameter of one tracking inflammatory acne lesion will be performed by a dermatologist using a skin ruler. The maximum diameter in millimeters (mm) will be recorded at each time point.
Clinical scoring for Cheek Sebaceous Pores | Timepoint 2Week before baseline, Baseline，Time point immediate, Time point at 1Week , Time point at 4Week, Time point at 5Week, Time point at 6Week.
  Clinical scoring for cheek sebaceous pores (based on the Skin Aging Atlas, Asian type), as well as for redness, smoothness, radiance, brightness, and softness, will be performed by a dermatologist using a visual grading scale from 0 to 9, as defined in the protocol. Half-point scores (e.g., 0.5) may be used.
Skin hydration on the cheeks | Baseline, Time point at 1Week , Time point at 4Week, Time point at 5Week, Time point at 6Week.
  Skin hydration on the cheeks will be measured by Corneometer® CM 825 by trained technician.
TEWL on the cheeks | Baseline, Time point at 1Week , Time point at 4Week, Time point at 5Week, Time point at 6Week.
  TEWL on the cheeks will be measured by Vapometer by trained technician.
Sebum secretion on forehead | Baseline, Time point at 1Week , Time point at 4Week, Time point at 5Week, Time point at 6Week.
  Sebum secretion on forehead will be measured by Sebumeter® SM 815 by trained technician.
Image capture and analysis（facial photo） | Baseline, Time point immediate, Time point at 1Day, Time point at 3Day, Time point at 1Week , Time point at 4Week, Time point at 5Week, Time point at 6Week.
  The facial photo will be captured by VISIA CRP (Canfield, Gen 5.0) on left, front and right sides with Standard 1, Cross-Polarized, Parallel-Polarized, UV operated by trained technician.
  -Demo for Pore area, skin reflection under Standard 1 and acne demo under Cross-Polarized.
One tracking active acne image | Baseline，Time point immediate, Time point at 1Day, Time point at 3Day, Time point at 1Week.
  One active inflammatory acne lesion will be imaged using Antera® 3D (Miravex). Image analysis will include acne volume (mm³) and area (mm²), using the Antera 3D CS software.
Image Capture and Analysis(RCM) | Baseline, Time point 4Week.
  RCM (Reflectance Confocal Microscopy) will be captured on target acne
  -microcomedone ratio, size, hyper-keratin ratio will be analyzed.
Image Capture using VisioScan® VC20plus | Baseline, Time point 4Week.
  Skin image will be captured using VisioScan® VC20plus (Courage + Khazaka) with Sebufix® F 16. Sebum production will be evaluated through sebum spot size and sebum distribution gradient using SELS software.

SECONDARY OUTCOMES:
Consumer Questionnaire | Time point immediate, Time point at 1Week , Time point at 4Week.
  Consumer-reported outcomes will be assessed using a self-assessment questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ping Xu, Master, Principal Investigator — Shanghai China-norm Quality Technical Service Co., Ltd.
Locations (1):
- Shanghai China-norm Quality Technical Service Co., Ltd., Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
This Data Sharing Plan (DSP) aims to promote the open exchange and reuse of de-identified individual participant data (IPD) from cosmetic clinical research, including study protocols, case report forms (CRFs), and statistical analysis plans (SAPs). The shared data will be made available through compliant platforms to eligible researchers in dermatology, cosmetic science, and related fields, following ethical principles and data protection regulations. Users must sign a Data Use Agreement (DUA) to ensure data security, privacy protection, and compliance with research purposes.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 18-Month Duration: The data sharing period starts upon study completion and PRS registration completion.
  Timeline:
  Months 2-3: Data de-identification, metadata preparation, and platform integration.
  Month 4: Official launch of data access.
Access Criteria: Primary Platform:
  ResMan (www.medresman.org.cn) - China's leading medical research data repository.
  Eligibility:
  Researchers/affiliates from academic institutions, hospitals, or registered research organizations.
  Engaged in dermatology, cosmetic science, or related fields. Able to demonstrate ethical compliance and data security capabilities.
URL: http://www.medresman.org.cn